CLINICAL TRIAL: NCT00320723
Title: Nicotine Replacement Therapy Added to Cognitive Behavioral Therapy for Smoking Cessation in Patients With Major Mental Illness
Brief Title: Nicotine Replacement Therapy for Smoking Cessation in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Responsible Party: A Eden Evins, MD, MPH, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMH CORRC 20-01
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; smoking cessation; nicotine; patch; bupropion; nicotine replacement therapy; cognitive behavioral therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Smoking Cessation | interventions — Bupropion; Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: bupropion, transdermal nicotine patch

SUMMARY:
This proposal seeks to evaluate a pilot smoking cessation treatment program that will combine nicotine replacement therapy with or without bupropion sustained-release (SR) with cognitive behavioral therapy for smoking cessation in patients with major mental illness.

DETAILED DESCRIPTION:
Background:

Seventy-four to 92% of patients with schizophrenia smoke cigarettes compared to 24% of the adult US population and 18% of adults in Massachusetts (1-3). Patients with schizophrenia also smoke more cigarettes on average per day (4) and attain higher serum levels of cotinine, the primary metabolite of nicotine, a finding attributed to deeper smoke inhalation (5). Cigarette smoking has been identified as the single most important source of preventable morbidity and premature mortality in the general U.S. population for the last 29 years (6, 7). Compounded by the problem that patients with schizophrenia live a less healthy lifestyle (8) and may be less likely to receive adequate routine and preventative medical care (9-12), heavy smoking represents a significant and neglected public health problem for people with schizophrenia. Patients with schizophrenia clearly have greater morbidity and early mortality from 'natural causes' than people without schizophrenia (13-22) and are more likely to die prematurely from cardiovascular or pulmonary disease (14, 19, 23-26). Women with schizophrenia have been shown to have increased risk of premature death from cancer (24) and previous studies showing lower mortality from cancer in patients with schizophrenia compared to the general population have not been confirmed (14, 27, 28). Successful smoking cessation programs for patients with schizophrenia could reduce this increased medical morbidity and mortality. A recent report of patterns of nicotine use in a cohort of 50 patients with schizophrenia or schizoaffective disorder underscores this point: the cohort had a mean age of 47 years and mean age at onset of daily smoking of 20 years; 45.8% reported they currently have a smoking related health problem; 95.8% had tried unsuccessfully to cut down on their smoking; 70% had made a serious attempt to quit smoking (29). Smoking cessation programs for patients with schizophrenia have reported compliance rates as high as 80% (30).

Nicotinic receptors have been shown to be reduced in number in patients with schizophrenia (31, 32) and heavy smoking in schizophrenia may be attributable to attempts to overcome this deficit. Benefits of nicotine to patients with schizophrenia include reversal of some of the specific cognitive deficits associated with schizophrenia and antipsychotic treatment [(33-37). Nicotine has been shown to improve learning, visual and spatial working memory, attention, auditory sensory gating smooth pursuit eye movements and reaction time (38, 39). The positive effects of chronic nicotine treatment appear to persist over time, and in some studies, improvements in cognition with chronic nicotine treatment become more robust over time (40). Smoking cessation in patients with schizophrenia is associated with increase in positive symptoms (30). Treatment with atypical antipsychotics may enhance the effectiveness of smoking cessation treatment (41-43). The mechanism of this effect is not known but may be due to decreased extrapyramidal side effects, improved efficacy for negative symptoms or effects on glutamatergic systems. Combination of NRT and antidepressant medication has been shown to increase cessation rates over monotherapy with NRT (44) but not over antidepressant medication alone (45).

Nicotine replacement therapy (NRT) is a powerful aid to smoking cessation with well established efficacy (46-49) in non-psychiatric patients and has been proposed as a potential tool in increasing smoking harm reduction in persons unable to achieve smoking abstinence (50). Smoking cessation outcomes in patients with schizophrenia using NRT have been extremely variable. Ziedonis and colleagues used a range of doses of NRT administered by patch, gum or combination in addition to CBT for up to 10 weeks in 24 patients with schizophrenia (51). Twelve subjects completed the trial. The cessation rate was 13% at 6 months (51). In one study, atypical antipsychotic agents, in combination with the nicotine transdermal patch, have been shown to significantly enhance the rate of smoking cessation (55.6% in the atypical agent group versus 22.2% in the typical group) (41). In this study the overall end of treatment point prevalence smoking cessation rate in 45 patients with schizophrenia was 35%. In another study of the acute effects of transdermal nicotine patch in psychiatric patients, however, no patients quit smoking acutely, and only heavy smokers reduced their cigarette consumption (52).

Safety of NRT in patients with schizophrenia has only been evaluated on a very small scale. One important trial examined the effects of a 21 mg nicotine patch on smoking behavior, nicotine levels in blood and signs of toxicity in patients with schizophrenia (53). In this crossover trial, 10 male veterans were monitored while wearing nicotine vs placebo patches. The nicotine patch condition was associated with increased nicotine levels without signs of toxicity and decreased CO levels in 80% of patients. No trials have reported worsening of psychiatric symptoms with NRT. Larger studies in which NRT is combined with behavioral support are needed to evaluate the efficacy and safety of NRT in schizophrenia.

Treatment Component:

Subjects will be outpatients who are clinically stable and currently in treatment for schizophrenia or schizoaffective disorder. Subjects will be recruited through referral from case managers, residential treatment settings and outpatient treaters. Subjects must smoke =1/2 pack per day of cigarettes and wish to quit smoking.

Subjects will be randomly assigned to receive cognitive behavioral smoking cessation therapy CBT) with nicotine patch (NRT) plus placebo or nicotine patch combined with bupropion SR. Subjects who are unable to tolerate or who have a contraindication to treatment with zyban may be enrolled to receive CBT and open label NRT alone. All subjects will receive a 12 session group cognitive behavioral therapy (CBT) program designed for smoking cessation treatment in patients with schizophrenia in addition to pharmacologic treatment.

Evaluation Component:

The evaluation component of this protocol involves monitoring patients for stability of psychiatric symptoms, serum levels of psychiatric medications, and medication side effects at baseline and weeks 4, 8, 12 and 14 and degree of smoking reduction or cessation weekly during the treatment intervention and at 6, 12 and 24 months.

At baseline, subjects will complete a demographic questionnaire. Prior to beginning treatment, subjects will be evaluated for symptoms of psychosis, depression, anxiety, and medication side effects with standard clinical rating scales that include the schedule for assessment of negative symptoms (SANS), positive and negative symptom scale (PANSS), Hamilton depression scale (HamD), Hamilton anxiety scale (HamA), abnormal involuntary movement scale (AIMS), Simpson Angus Scale, and SAFTEE. A brief cognitive battery will include tests of response inhibition (the single trial Stroop), vigilance (continuous performance test), verbal fluency (FAS), verbal memory (California Verbal Learning Test), working memory (letter number span), non-verbal memory (Benton visual retention test), psychomotor ability (grooved peg board task), and executive functioning (trail making or tower of London). Baseline carbon monoxide (CO) measurements will be used with self report to verify number of cigarettes smoked per day. Serum will be drawn for cotinine and antipsychotic levels at baseline. Weight will be checked at baseline, 12 and 24 weeks.

Subjects will set a quit date between weeks 3 and 4. The evaluation battery will be repeated at week 4 just following the quit date. It will also be repeated at week 12 when patients discontinue the group and medication treatment. An evaluation that includes the clinical battery and CO measurement will be performed at week 14, two weeks following termination of smoking cessation treatment and at week 24. Subjects will also be contacted at 1 and 2 years for follow up self report of tobacco use and CO measurement.

Specific Aims: Treatment

1. Increase availability of nicotine replacement therapy, which is not currently available by prescription, to patients with major mental illness.
2. Train staff members with expertise in treating patients with major mental illness to be Tobacco Treatment Specialists using the training protocol developed by University of Massachusetts Medical School in collaboration with the Massachusetts Department of Public Health.
3. Establish a network of centers able to deliver tobacco treatment to patients with major mental illness.

Specific Aims: Evaluation

1. Evaluate smoking cessation rates, smoking reduction rates and stability of psychiatric symptoms in patients with schizophrenia and schizoaffective disorder during a smoking cessation attempt using cognitive behavioral therapy combined with NRT plus placebo and NRT + bupropion SR.
2. Evaluate safety of nicotine replacement therapy in patients with schizophrenia and schizoaffective disorder when combined with antipsychotic medications.
3. Evaluate safety of nicotine replacement therapy in patients with schizophrenia and schizoaffective disorder when combined with bupropion SR and antipsychotic medications.

Hypotheses:

1. Nicotine replacement therapy combined with bupropion SR and cognitive behavioral therapy will be associated with improvement in smoking cessation and smoking reduction rates when compared to NRT alone added to CBT in patients with schizophrenia and schizoaffective disorder.
2. Nicotine replacement therapy combined with bupropion SR will be associated with improvement in negative symptoms, depression and impulsivity when compared to NRT alone in patients with schizophrenia and schizoaffective disorder who quit smoking.
3. Concurrent treatment with atypical antipsychotic medications will further enhance the effectiveness of NRT combined with bupropion SR and NRT plus placebo for smoking cessation and reduction in patients with schizophrenia and schizoaffective disorder compared to concurrent treatment with conventional antipsychotics.
4. Patients with low baseline cotinine = 250 ng/ml will have higher cessation rates than patients with high baseline cotinine >250 ng/ml.

ELIGIBILITY:
Inclusion Criteria

1. Women and men aged 18-70 with a diagnosis of schizophrenia or schizoaffective disorder (depressed type or bipolar type) by structured diagnostic interview or chart review
2. Clinically stable on a stable dose of antipsychotic medication for at least one month, no current active suicidal ideation
3. Expired air CO > 9 ppm and self report of smoking >1/2 pack per day of cigarettes
4. Willing to set a smoking quit date within one month of beginning treatment
5. Not treated with investigational medication in the past 30 days
6. Competent to provide informed consent or able to provide assent with legal guardian informed consent
7. Meet DSM-IV criteria for Nicotine Dependence, as determined with the Fagerstrom Nicotine Tolerance Questionnaire (FTQ) (Fagerstrom, 1978)
8. Compliant with last 3 clinic visits

Exclusion Criteria

1. Diagnosis of dementia, neurodegenerative disease, current anorexia/bulimia nervosa, current substance abuse or dependence disorders, including alcohol, active within the last 3 months or any Axis I DSM-IV diagnosis other than schizophrenia or schizoaffective disorder
2. Severe or unstable angina; myocardial infarction in the past 2 weeks; untreated peptic ulcer; life-threatening arrhythmia; poorly controlled insulin dependent diabetes mellitus, uncontrolled hypertension, cerebrovascular event within six months; or allergy to a nicotine patch. Serious illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease that is not stabilized such that hospitalization for treatment of that illness is likely within the next two months
3. Patients who, in the investigator's opinion, pose a current severe homicide or suicide risk
4. Subjects with a history of skin diseases (e.g., psoriasis), skin allergies, or strong reactions to topical preparations, medical dressings or tapes
5. Current use of topical medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-07; Study Completion 2005-12

PRIMARY OUTCOMES:
improvement in smoking cessation and smoking reduction rates when compared to NRT alone added to CBT in patients with schizophrenia and schizoaffective disorder

SECONDARY OUTCOMES:
improvement in negative symptoms, depression and impulsivity when compared to NRT alone in patients with schizophrenia and schizoaffective disorder who quit smoking

CONTACTS AND LOCATIONS:
Overall Officials: A Eden Evins, MD, MPH, Principal Investigator — North Suffolk Mental Health Association
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States